CLINICAL TRIAL: NCT05581706
Title: The Effects of Calcium Hydroxide and Double Antibiotic Paste on Radiographic Outcomes and Periapical MMP-8 Levels in Regenerative Endodontic Procedures: A Randomized Clinical Trial
Brief Title: Regenerative Endodontics Using Different Intracanal Medicaments on Radiographic Outcomes and Periapical MMP-8 Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Burç Pekpınarlı, Principal investigator, Asst. Dr, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Regenerative Endodontics
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Regenerative Endodontics
Keywords: regenerative endodontics; intracanal medicaments; MMP-8
MeSH Terms: interventions — Specimen Handling; Fluoroimmunoassay

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Regenerative endodontic treatment with calcium hydroxide (Active Comparator): Regenerative endodontic treatment (RET) performed with procedures of American Association of Endodontics (AAE) in two sessions. At the end of the first session, periapical tissue fluid samples (baseline samples) were collected.
  Calcium hydroxide medicament was prepared by mixing with sterile distilled water and then placed in the coronal 1/3 of the root canals.
  In the second session (14 days after first treatment), the medicaments in the root canals were carefully removed with 5 ml sterile distilled water irrigation. Periapical tissue fluid samples were obtained from the distal canal using the same protocol as described previously (final samples). Then RET was finished according to the treatment protocol of AAE.
  Interventions: Combination Product: Place the freshly prepared calcium hydroxide in to the root canals
- Regenerative endodontic treatment with double antibiotic paste (Active Comparator): Regenerative endodontic treatment (RET) performed with procedures of American Association of Endodontics (AAE) in two sessions. At the end of the first session, periapical tissue fluid samples (baseline samples) were collected.
  Double antibiotic paste (DAP) was prepared by mixing same amount of metronidazole and ciprofloxacin powdered antibiotics (1:1) and combined with sterile distilled water to form an ointment. DAP was introduced in roots canals using a lentulo to fill the entire root canal space.
  In the second session (14 days after first treatment) after removal of DAP in the root canals, periapical tissue fluid samples were obtained the same protocol as described previously (final samples). Then RET was finished according to the treatment protocol of AAE.
  Interventions: Combination Product: Place the freshly prepared double antibiotic paste in to the root canals
- Radiographic evaluation (Active Comparator): Pre-operative, post-operative and final recall (12th months follow up) standart digital radiographs were taken from patients with film holder. The radiographs saved and transferred to Image J software (version 1.47, National Institutes of Health, Bethesda, MD). The standardized radiographs were further aligned using the TurboReg plugin (Biomedical Imaging Group, Swiss Federal Institute of Technology, Lausanne, Switzerland) within the Image J toolkit to minimize any distortions caused by variability in the angulation.
  All images were calibrated according to size #2 SPP (vertical dimension 31 mm, horizontal dimension 41 mm) using the ''set scale'' option in Image J. Thereafter, the root lengths, root width and radiographic root area were measured on both preoperative and final recall images to evaluate treatment outcomes.
  Interventions: Diagnostic Test: Taking standart periapical radiography with film holder
- Periapical tissue exudate sample collection and Immunofluorometric assay MMP-8 (Active Comparator): At the end of the first session, periapical tissue fluid samples (baseline samples) were collected by introducing 3 sterile #45 paper points into the root canal until 2 mm passing through the root apex from the distal canal. After waiting for 1 min, the paper points were withdrawn, the tip was cut from 4 mm and were transferred to sterile Eppendorf tubes. At the beginnign of the second session periapical tissue fluid samples were obtained from the distal canal using the same protocol as described in the first session (final samples).
  Baseline and final MMP-8 concentrations were determined by a time-resolved immunofluorometric assay (IFMA). The monoclonal MMP-8 specific antibodies 8708 and 8706 (Oy Medix Biochemica Ab, Espoo, Finland) were used as a catching antibody and a tracer antibody, respectively. The tracer antibody was labeled using europium-chelate
  Interventions: Other: Sample collection for immunofluorometric assay

INTERVENTIONS:
Combination Product: Place the freshly prepared calcium hydroxide in to the root canals — Calcium hydroxide (Merck, Darmstadt, Germany): prepared by mixing with sterile distilled water and then placed in the coronal 1/3 of the root canals.
  Other Names: Ca(OH)2 medicament
  Arms: Regenerative endodontic treatment with calcium hydroxide
Combination Product: Place the freshly prepared double antibiotic paste in to the root canals — Double antibiotic paste (DAP): metronidazole (Flagyl, Sanofi-Aventis, Turkey) and ciprofloxacin (Cipro, Biofarma, Turkey) powdered antibiotics were stored and sealed in airtight containers. The same amount of each drug powder (1:1) was mixed and the mixed samples were combined with sterile distilled water to form an ointment. DAP was introduced in roots canals using a lentulo to fill the entire root canal space.
  Other Names: DAP medicament
  Arms: Regenerative endodontic treatment with double antibiotic paste
Diagnostic Test: Taking standart periapical radiography with film holder — Post-operative periapical radiographs were obtained with Digora Optime SPP system (Soredex Corp., Tuusula, Finland) using intraoral film holders to keep the plates parallel to the long axis of the teeth. A size #2 SPP was used for all exposures. SPPs were exposed with a Gendex Oralix DC dental x-ray unit (Gendex Dental Systems, Milan, Italy) operating at 60 kVp, 7 mA, 0.25 sec. and the plates were scanned immediately after exposure. The clinical and radiographical follow up was performed on 12th months.
  Image-J program (version 1.47, National Institutes of Health, Bethesda, MD) with TurboReg plug-in (Biomedical Imaging Group, Swiss Federal Institute of Technology, Lausanne, Switzerland) was used to determine the increase in root length, root width, and radiographic root area at 12th month follow up.
  Other Names: Determination of rooth lenght, rooth width, radiographic root area
  Arms: Radiographic evaluation
Other: Sample collection for immunofluorometric assay — Periapical exudate samples were collected at the beginning of the RET and at 14th day. MMP-8 levels were measured by immunofluorometric assay (IFMA). Briefly, two monoclonal MMP-8-specific antibodies, 8708 and 8706 (Oy Medix Biochemica Ab, Espoo, Finland) were used as catching antibody and tracer antibody, respectively. Samples were diluted in enzyme buffer (50 mM Tris-HCl, pH 7.5; 0.2 mM NaCl, 1 mM CaCl2). Twenty microlitres of samples and 80 μl of assay buffer (20 mM Tris-HCl, pH 7.5, 0.5 M NaCl, 5 mM CaCl2, 0.5% BSA, 0.05% sodium azide and 20 mg/l diethylenetriaminepentaacetic acid with 2 μg/ml normal mouse serum) were pipetted into the wells. The tracer antibody was labelled using europium chelate. After adding the enhancement solution, fluorescence was measured using a 1234 Delfia Research Fluorometer (Wallac, Turku, Finland).
  Other Names: IFMA
  Arms: Periapical tissue exudate sample collection and Immunofluorometric assay MMP-8

SUMMARY:
Two-session regenerative endodontic treatment was applied to 20 immature mandibular first molars with symptomatic irreversible pulpitis and symptomatic apical periodontitis. At the end of the first session, calcium hydroxide [Ca(OH)2] was applied to 10 randomly selected teeth and double antibiotic paste (DAP) intracanal medicaments were applied to the other 10 teeth. The effects of intracanal medicaments on periapical MMP-8 levels were determined by immunofluorometric assay (IFMA) in periapical tissue fluid samples taken from the distal root canal in the first and second sessions.

DETAILED DESCRIPTION:
The aim of the study was to investigate the effects of two different intracanal medicaments used during regenerative endodontic treatment (RET) on periapical MMP-8 in relation to the radiological outcomes of RET. After local anesthesia and rubber dam isolation were provided, disinfection procedures were applied gently in accordance with the current RET protocol of American Association of Endodontics (AAE) on the molar teeth. Periapical tissue fluid samples were taken with paper points placed to protrude 2 mm from the distal root canal tip. Calcium hydroxide [Ca(OH)2] was placed in 10 randomly selected teeth and double antibiotic paste (DAP) intracanal medicaments were placed in the other 10 teeth. Fourteen days later in the second session, the final sampling procedure was performed as in the first session. Then, the treatment was completed according to the current RET protocol of AAE and permanent restorations were made. The success of the treatment and its effect on root development were evaluated by comparing the standard radiographs taken at the end of the treatment and 12 months follow up. MMP-8 levels were measured by immunofluorometric assay (IFMA) in the periapical tissue fluid samples. First and second session MMP-8 levels were compared according to the groups of medicaments [Ca(OH)2 and DAP groups] placed in the root canals.

ELIGIBILITY:
Inclusion Criteria:

- Healthy children with irreversible pulpitis with symptomatic apical periodontitis (SIP-SAP), indication for RET and informed consent from the patients.

Exclusion Criteria:

* Children with extra oral swelling or luxation with a deep periodontal pocket and whom application of RET was contraindicated.
* The teeth were indicated for vital pulp therapy (assesed during treatment)
* Children who have used antibiotics in the past 3 months and are uncooperative during treatment
* Children who have used any painkillers during the treatment

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical healing according to presence of clinical symptoms | 12 months
  All patients were called for follow up visits. The clinical healing was determined by examining clinical symptoms including presence of pain, tenderness to percussion and palpation, presence of sinus tract or swelling, and mobility. All teeth were asymptomatic at follow up appointments. If one of these symptoms occurred, it could considered as failure.
Periapical healing according to change in amount of root hard tissues | 12 months
  All periapical radiolucency detected due to apical periodontitis were healed. Significant increases in radiographic root length, root width and RRA was observed at 12th month.
MMP-8 levels from periapical tissue fluid samples | 14 day
  There was a statistically significant increase in MMP-8 levels on day 14 compared to baseline in both Ca(OH)2 and DAP groups. The increase in MMP-8 levels was higher in the DAP group compared to Ca(OH)2 group, however no statistically significant difference was observed between 2 groups regarding the final (14th day) MMP-8 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Burç Pekpınarlı, Principal Investigator — Ege University Faculty of Dentistry
Locations (1):
- Ege University Faculty of Dentistry Pediatric Dentistry, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torabinejad M, Alexander A, Vahdati SA, Grandhi A, Baylink D, Shabahang S. Effect of Residual Dental Pulp Tissue on Regeneration of Dentin-pulp Complex: An In Vivo Investigation. J Endod. 2018 Dec;44(12):1796-1801. doi: 10.1016/j.joen.2018.09.005. PMID 30477665
- [Background] Sabeti M, Golchert K, Torabinejad M. Regeneration of Pulp-Dentin Complex in a Tooth with Symptomatic Irreversible Pulpitis and Open Apex Using Regenerative Endodontic Procedures. J Endod. 2021 Feb;47(2):247-252. doi: 10.1016/j.joen.2020.09.021. Epub 2020 Oct 10. PMID 33045267
- [Background] Wahlgren J, Salo T, Teronen O, Luoto H, Sorsa T, Tjaderhane L. Matrix metalloproteinase-8 (MMP-8) in pulpal and periapical inflammation and periapical root-canal exudates. Int Endod J. 2002 Nov;35(11):897-904. doi: 10.1046/j.1365-2591.2002.00587.x. PMID 12453017
- [Background] Kuula H, Salo T, Pirila E, Tuomainen AM, Jauhiainen M, Uitto VJ, Tjaderhane L, Pussinen PJ, Sorsa T. Local and systemic responses in matrix metalloproteinase 8-deficient mice during Porphyromonas gingivalis-induced periodontitis. Infect Immun. 2009 Feb;77(2):850-9. doi: 10.1128/IAI.00873-08. Epub 2008 Nov 24. PMID 19029300
- [Background] Bose R, Nummikoski P, Hargreaves K. A retrospective evaluation of radiographic outcomes in immature teeth with necrotic root canal systems treated with regenerative endodontic procedures. J Endod. 2009 Oct;35(10):1343-9. doi: 10.1016/j.joen.2009.06.021. Epub 2009 Aug 15. PMID 19801227
- [Background] Reynaud af Geijersstam A, Sorsa T, Stackelberg S, Tervahartiala T, Haapasalo M. Effect of E. faecalis on the release of serine proteases elastase and cathepsin G, and collagenase-2 (MMP-8) by human polymorphonuclear leukocytes (PMNs). Int Endod J. 2005 Sep;38(9):667-77. doi: 10.1111/j.1365-2591.2005.01011.x. PMID 16104981
- [Background] Martinho FC, Nascimento GG, Leite FR, Gomes AP, Freitas LF, Camoes IC. Clinical influence of different intracanal medications on Th1-type and Th2-type cytokine responses in apical periodontitis. J Endod. 2015 Feb;41(2):169-75. doi: 10.1016/j.joen.2014.09.028. Epub 2014 Nov 11. PMID 25453567
- [Derived] Pekpinarli B, Kaval ME, Cogulu D, Ilhan B, Sorsa T, Tervahartiala T, Oncag O. The effect of calcium hydroxide and double antibiotic paste on radiographic outcomes and periapical MMP-8 levels in regenerative endodontic procedures: a randomized clinical trial. J Appl Oral Sci. 2024 Sep 20;32:e20240122. doi: 10.1590/1678-7757-2024-0122. eCollection 2024. PMID 39319904